CLINICAL TRIAL: NCT01060514
Title: Phase I Study of Pazopanib in Combination With Vinorelbine in Patients With Metastatic Non-Small Cell Lung Cancer (NSCLC) and Breast Cancer
Brief Title: Pazopanib + Vinorelbine in Non Small Cell Lung Cancer (NSCLC) and Breast Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of timely accrual.
Sponsor: Northwestern University (Other)
Collaborators: Robert H. Lurie Cancer Center (Other)
Responsible Party: Principal Investigator, Jyoti Patel, Principal Investigator, Northwestern University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NU 09L1; STU00019948 (Other: Northwestern University IRB); NCI-2010-01850 (Other: NCI CTRP#)
Record Dates: First submitted 2010-01-29; First posted 2010-02-02 (Estimated); Last update posted 2013-10-30 (Estimated); Status verified 2013-10

CONDITIONS: Metastatic Non Small Cell Lung Cancer; Metastatic Breast Cancer
Keywords: Lung cancer; Breast cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Breast Neoplasms; Lung Neoplasms | interventions — pazopanib; Vinorelbine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pazopanib + Vinorelbine (Experimental)
  Interventions: Drug: Pazopanib; Drug: Vinorelbine

INTERVENTIONS:
Drug: Pazopanib — dose escalation, administered orally, daily
Drug: Vinorelbine — dose escalation, IV days 1 and 8 of every cycle (cycles begin every 3 weeks)
  Other Names: Navelbine

SUMMARY:
The purpose of this study is to determine the highest dose of Vinorelbine and Pazopanib that can be given together without causing severe side effects. Also, this study will evaluate what effects (good and bad) that the treatment has on patients and their cancer.

DETAILED DESCRIPTION:
This study involves an investigational drug called pazopanib in combination with the chemotherapy drug vinorelbine. An investigational drug is a drug that has not been approved by the U.S. Food and Drug Administration (FDA) for use in the United States. Vinorelbine has been FDA approved to treat patients with NSCLC and breast cancer. Pazopanib is a vascular endothelial growth factor inhibitor, which means it may prevent the tumor from growing its own blood vessels thereby interfering with the growth of the tumor. Participants in this study will be assigned to one of three groups with each group receiving a higher dose of vinorelbine and pazopanib than the previous group. Vinorelbine will be given through a needle in the vein on days 1 and 8 of each 21 day study treatment cycle. Pazopanib is a pill which will be taken by mouth every day during the 21 day study treatment cycle.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Patients must have diagnosis of breast cancer or non small cell lung cancer
* Patients must have evaluable disease
* Women of childbearing potential and sexually active males must commit to the use of effective contraception while on study.
* Patients must have given signed, informed consent prior to registration on study.

Exclusion Criteria:

* Patients must not be pregnant and/or lactating.
* Patients must not be receiving any other investigational agents.
* No prior exposure to vinorelbine or other VEGF inhibitors as treatment for metastatic disease
* Patients must not have received prior therapy (including radiation, surgery, and/or chemotherapy) within 30 days
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to pazopanib or vinorelbine.
* Patients cannot have received more than 2 prior chemotherapy regimens for lung cancer or 3 prior chemotherapy regimens for breast cancer. This criterion can be discussed further with the study doctor.
* Must not have uncontrolled illness including, but not limited to: ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmic, psychiatric illness/social situations that would limit compliance with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2010-02; Primary Completion 2012-02 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose (MTD), and the recommended Phase II dose to be used in patients with metastatic NSCLC and breast cancer. | at study completion (estimated at 2 years)

SECONDARY OUTCOMES:
To determine the response rate, progression free survival and overall survival in patients with metastatic NSCLC and metastatic breast cancer treated with pazopanib in combination with vinorelbine. | imaging done every 6 weeks
To characterize dose limiting toxicities (DLT). | labs drawn weekly
To determine the pharmacokinetic effect of pazopanib on vinorelbine. | labs drawn on days 1 and 22

CONTACTS AND LOCATIONS:
Overall Officials: Jyoti D Patel, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Northwestern Medical Faculty Foundation, Chicago, Illinois, United States